CLINICAL TRIAL: NCT01888380
Title: Post-mortem Cross-sectional Imaging With Guided Biopsy; A Comparative Study With Conventional Autopsy in Foetuses, Neonates, Infants and Children
Brief Title: The Paediatric Virtual Autopsy Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: Paediatric virtopsy
Record Dates: First submitted 2013-06-17; First posted 2013-06-27 (Estimated); Last update posted 2021-01-11 (Actual); Status verified 2020-03

CONDITIONS: Stillbirth; Newborn Death; Sudden Infant Death
Keywords: Autopsy; Minimally invasive; Foetuses; Newborns; Children; Adolescents
MeSH Terms: conditions — Stillbirth; Perinatal Death; Sudden Infant Death | interventions — Autopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Foetuses (Experimental): * still birth and termination of pregnancies
  * intervention: minimally invasive, virtual autopsy
  Interventions: Procedure: Minimally invasive, virtual autopsy; Procedure: Conventional autopsy
- Newborns (Experimental): * who died of natural- and non-natural cause
  * intervention: minimally invasive, virtual autopsy
  Interventions: Procedure: Minimally invasive, virtual autopsy; Procedure: Conventional autopsy
- Children and adolescents (Experimental): * who died of natural- and non-natural cause
  * intervention: minimally invasive, virtual autopsy
  Interventions: Procedure: Minimally invasive, virtual autopsy; Procedure: Conventional autopsy

INTERVENTIONS:
Procedure: Minimally invasive, virtual autopsy — Post-mortem cross-sectional imaging with CT-guided biopsy
  Other Names: Virtopsy
Procedure: Conventional autopsy
  Other Names: Postmortem

SUMMARY:
In light of declining autopsy rates around the world, post-mortem MR imaging is a promising alternative to conventional autopsy in the investigation of infant death. A major drawback of this non-invasive autopsy approach is the fact that histopathological and microbiological examination of the tissue is not possible. The objective of this prospective study is to compare the performance of minimally invasive, virtual autopsy, including CT-guided biopsy, with conventional autopsy procedures in a paediatric population.

Foetuses, newborns, infants and children that are referred for autopsy at three different institutions associated with the University of Zurich will be eligible for recruitment. All bodies will be examined with a commercial CT and a 3 Tesla MRI scanner, and investigators will be blinded to the results of conventional autopsy. After cross-sectional imaging, CT-guided tissue sampling will be performed by a multifunctional robotic system (Virtobot) allowing for automated post-mortem biopsies. Virtual autopsy results will be classified with regards to the likely final diagnosis and major pathological findings and compared to the results of conventional autopsy, which remains the diagnostic gold standard.

This interdisciplinary study will determine whether virtual autopsy will narrow the gap in information between non-invasive and traditional autopsy procedures.

ELIGIBILITY:
Inclusion criteria:

* Stillborn infants ≥ 16 0/7 weeks of gestational age (GA)
* Live born infants ≥ 16 0/7 weeks GA until adolescents up to 16 years of age, who died of natural- and non-natural cause (trauma, homicide, suicide and intoxication).

Exclusion criteria:

* Deceased infants who are donors of organs
* Lack of parental consent

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 105 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Percentage of cases for which virtual autopsy correctly identifies the cause of death and/or major pathological lesions | 8 weeks
  The diagnoses established in both ways by the two independent teams will be compared, the autopsy results being the gold standard. The primary outcome will be the percentage of cases for which virtual autopsy correctly identifies the diagnostic category.

SECONDARY OUTCOMES:
Clinical indication | 8 weeks
  Number of false positive and false negative results of virtual autopsy will be calculated for each organ system.
MR Protocol | 8 weeks
  To optimize a protocol for MR imaging examinations in deceased foetuses, neonates, infants and children
Change in the ante-mortem diagnosis | 8 weeks
  The proportion of cases, for which virtual autopsy leaded to a change in ante-mortem diagnosis, will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Hans Ulrich Bucher, MD, Prof, Study Director — University Hospital Zurich, Division of Neonatology; Christoph Rüegger, MD, Principal Investigator — University Hospital Zurich, Division of Neonatology
Locations (4):
- Switzerland (4):
  - University Hospital Zurich, Division of Neonatology, Zurich, Canton of Zurich
  - Division of obstetrics, University Hospital Zurich, Zurich
  - University Children's Hospital Zurich, Zurich
  - Zurich Institute for Forensic Medicine, Zurich

REFERENCES:
- [Derived] Ruegger CM, Gascho D, Bode PK, Bruder E, Haslinger C, Ross S, Schmid K, Knopfli C, Hofer LJ, Held L, Martinez RM, Bucher HU; Virtopsy Study Group. Post-mortem magnetic resonance imaging with computed tomography-guided biopsy for foetuses and infants: a prospective, multicentre, cross-sectional study. BMC Pediatr. 2022 Aug 3;22(1):464. doi: 10.1186/s12887-022-03519-4. PMID 35918685
- [Derived] Ruegger CM, Bartsch C, Martinez RM, Ross S, Bolliger SA, Koller B, Held L, Bruder E, Bode PK, Caduff R, Frey B, Schaffer L, Bucher HU. Minimally invasive, imaging guided virtual autopsy compared to conventional autopsy in foetal, newborn and infant cases: study protocol for the paediatric virtual autopsy trial. BMC Pediatr. 2014 Jan 20;14:15. doi: 10.1186/1471-2431-14-15. PMID 24438163